CLINICAL TRIAL: NCT06380244
Title: Opioid-free Anesthesia as an Alternative to General Anesthesia in Abdominal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Tomasz Skladzien, MD PHD, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1072.6120.136.2023
Record Dates: First submitted 2024-04-16; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Analgesics, Opioid; Anesthesia, Endotracheal; Anesthesia, General
MeSH Terms: interventions — Anesthesia; Analgesics, Opioid

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid (No Intervention): general anesthesia (using remifentanil infusion intraoperatively). Standard monitoring during anaesthesia included arterial oxygen saturation, ECG, and non-invasive arterial blood pressure. Premedication was not used. The standard anaesthesia consisted of propofol (1.5-2 mg / kg body weight iv) and for induction. Infusion of remifentanil in a plasma target control infusion with a calculated plasma level of 1-6 ng/ml. Rocuronium (0.6 mg / kg body weight iv) was administered prior to intubation. AThe painkillers used would be metamizole, acetaminophen and oxycodone.
- OFA (Experimental): completely anesthetized without opioids (infusion of Ketamine, Lignocaine and Dexmedetomidine. Standard monitoring during anaesthesia included arterial oxygen saturation, ECG, and non-invasive arterial blood pressure. Premedication was not used. The standard anaesthesia consisted of propofol (1.5-2 mg / kg body weight iv) and for induction. Rocuronium (0.6 mg / kg body weight iv) was administered prior to intubation. The painkillers used would be metamizole, acetaminophen and oxycodone.
  Interventions: Other: anesthesia without opioids

INTERVENTIONS:
Other: anesthesia without opioids — Opioid free general anesthesia
  Arms: OFA

SUMMARY:
Due to the increasing number of reports of cancer progression in people undergoing surgery under general anesthesia using opioids, OFA is believed to have a favorable long-term prognostic effect, especially in cancer patients. The opioid-free protocol is also used in postoperative analgesia. It is estimated that up to 75% of surgical patients experience chronic postoperative pain, which has a particularly negative impact on the quality of life.

The investigators would like to compare pain during the first 48 postoperative hours of patients undergoing abdominal surgery who would be anesthetized with opioids and without opioids (patients would be randomly assigned to a group) (1, 2, 6, 12, 24 and 48 h after operations). A secondary objective will be to measure total oxycodone consumption in the postoperative period in both groups. Other secondary objectives: assessment of postoperative nausea and vomiting (PONV).

DETAILED DESCRIPTION:
All subsequent patients undergoing abdominal surgery will be randomly divided into two groups: one under completely opioid-free anesthesia (infusion of Ketamine, Lignocaine and Dexmedetomidine and inhalation of Desflurane) and the other group under combined general anesthesia (using an infusion of remifentanil intraoperatively). In the postoperative period, all patients will receive Oxycodone in a PCA pump or in the form of oral tablets [naloxone (naloxone hydrochloride) + oxycodone (oxycodone hydrochloride)] and co-analgesics in the form of Paracetamol and Metamizole. Opioid-free general anesthesia is a recognized method used during anesthesia. It allows participants to effectively control pain, reducing the number of complications associated with taking large doses of opioid drugs. It should be emphasized that it is approved for use in routine anesthetic practice, and whether such a technique will be used in a given patient depends only on the experience, knowledge and preferences of the anesthesiologist. It is used in everyday anesthetic practice, but there is no conclusive scientific data confirming its advantage in patients undergoing abdominal surgery, so currently it depends only on the individual experience, knowledge and preferences of the anesthesiologist whether such a technique will be used in a given patient.

Mulier et al. proposed an OFA scheme including the supply of dexmedetomidine, ketamine and lidocaine for the induction of anesthesia, which ensures sedation, analgesia and sympathomimetic therapy followed by simultaneous maintenance infusion of lidocaine and dexmedetomidine. The protocol proposed by Mulier et al. is widely used and accepted worldwide. Initially, it was used in patients undergoing bariatric procedures, and then for all types of surgical procedures.

In the postoperative period, patients will have their pain level assessed using the NRS scale 1, 2, 6, 12, 24 and 48 hours after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient's consent to participate in the study
* surgery within the abdominal cavity

Exclusion Criteria:

* patient's refusal to participate in the study
* inability to operate the PCA pump
* not understanding how the NRS scale works
* hypersensitivity to anesthetic drugs
* 1st or 2nd degree heart block.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain level | 2 days
  comparison of differences in pain levels. The numeric rating scale (NRS) will be used, it is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"

SECONDARY OUTCOMES:
Total long acting opioid consumption in oxycodone equivalents | 2 days
  the total dosage of given drug

CONTACTS AND LOCATIONS:
Locations (1):
- Jagiellonian University, Krakow, Lesser Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
We plan to share demografic data, type of surgery, score in NRS and opioid consumption dosage.
Supporting Information: Study Protocol
Time Frame: The data will be available in 2026 for 1 year